CLINICAL TRIAL: NCT04426188
Title: " Brain Changes After Repetitive Head Impacts in Soccer and the Effects of a Protective Device: Biomechanical, Cognitive, Electrophysiological and Multimodal Neuroimaging Study "
Brief Title: " Acute Brain Changes After Repetitive Headers in Soccer and the Effects of a Protective Device "
Acronym: Soccer-BRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2019/45
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Traumatic Brain Injury; Concussion, Brain
Keywords: Soccer; Traumatic Brain Injury; Heading; Acceleration; Neuroimaging; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Magnetic Resonance Imaging; Muscle Strength Dynamometer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without mouthguard (Sham Comparator): Heading series without mouthguard from machine-projected soccer balls at standardized speeds
  Interventions: Procedure: Heading series; Device: Magnetic Resonance Imaging (MRI); Other: Cognitive computerized assessment; Procedure: Electrophysiological records; Device: Dynamometer
- With mouthguard (Experimental): Heading series with mouthguard from machine-projected soccer balls at standardized speeds
  Interventions: Procedure: Heading series; Device: Magnetic Resonance Imaging (MRI); Other: Cognitive computerized assessment; Procedure: Electrophysiological records; Device: Dynamometer

INTERVENTIONS:
Procedure: Heading series — 10 headers from machine-projected soccer balls at standardized speeds
Device: Magnetic Resonance Imaging (MRI) — Brain MRI before and after a series
Other: Cognitive computerized assessment — Cognitive evaluation carried out with two computerized tools
Procedure: Electrophysiological records — Electrophysiological recording of Motor Evoked Potentials consisting of the application of transcranial magnetic stimulations (TMS) and the collection of muscle activity by electromyogram (EMG)
Device: Dynamometer — Measure of the strength of the neck muscles using a dynamometer

SUMMARY:
Soccer, the most popular sport in the world, exposes players to repeated head impacts and concussions, due to contact with another player or with the ground. Moreover, routine game-play in soccer involves intentional and repeated head impacts through ball "heading", with frequent high velocities, which might cause a transient brain dysfunction. In this pre-post prospective interventional study, 22 soccer players will perform 10 headers from machine-projected soccer balls at standardized speeds, modelling routine soccer practice. They will perform heading series in 2 different oral conditions, on different days at least 1 week apart: 1) Without mouthguard and tight jaws ; 2) With mouthguard and tight jaws. The strength of the neck muscles will be measured before the heading series. The kinematic of the movement will be recorded during each impact during the 2 heading series, as well as the activity of the jaw muscles which will be recorded by electromyogram. Before and after each heading series, electrophysiological data, multimodal magnetic resonance imaging (MRI), and cognitive computerized assessment will be acquired

ELIGIBILITY:
Inclusion Criteria:

Male 18 to 25 years, enrolled in French Social Security, recruited from the soccer teams of the University of Bordeaux

Exclusion Criteria:

* Abnormal neurological examination
* Taking drugs targeting the central nervous system
* Any unhealed injury
* History of head trauma, or other notion of central nervous system injury
* History of severe high blood pressure, diabetes, chronic cardiovascular pathology, progressive or debilitating disease
* Family history of epilepsy
* Contraindication to MRI: head circumference> 60 - Claustrophobia - Pacemaker, Implantable Neurostimulation, Implantable Defibrillator - Cochlear Implants - Ocular or cerebral ferromagnetic foreign body - refusal to be informed of an anomaly detected with MRI
* Individuals under legal protection or unable of giving their informed consent

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Mean acceleration (m/s²) | Week 4
  Mean linear and rotational acceleration of the head
Mean acceleration (m/s²) | Week 6
  Mean linear and rotational acceleration of the head

SECONDARY OUTCOMES:
Period of cortical silence (milliseconds) | Week 4
  Corticomotor inhibition measured in milliseconds using transcranial magnetic stimulation and electromyographic recordings.
Period of cortical silence (milliseconds) | Week 6
  Corticomotor inhibition measured in milliseconds using transcranial magnetic stimulation and electromyographic recordings.
Normalized score | Week 4
  Normalized score (Z-score) on the subtests of the computerized cognitive battery
Normalized score | Week 6
  Normalized score (Z-score) on the subtests of the computerized cognitive battery
Average time | Week 4
  Average time on the subtests of the computerized cognitive battery
Average time | Week 6
  Average time on the subtests of the computerized cognitive battery
Mean strength ratio (Newton) | Week 4
  Mean strength ratio between flexor and extensor muscles of the neck measured in Newton using a dynamometer
Mean strength ratio (Newton) | Week 6
  Mean strength ratio between flexor and extensor muscles of the neck measured in Newton using a dynamometer
T-size measure | Week 4
  Functional connectivity at rest in MRI
T-size measure | Week 6
  Functional connectivity at rest in MRI

CONTACTS AND LOCATIONS:
Overall Officials: Hélène CASSOUDESALLE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France